CLINICAL TRIAL: NCT04096989
Title: The Development and Effectiveness of Traditional Chinese Medicine Regimen-based Lifestyle and Mobile Health Application Intervention for People With Prediabetes
Brief Title: The Effect of Traditional Chinese Medicine Regimen-based Lifestyle Mobile Health APP in Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08-X-026
Record Dates: First submitted 2019-09-10; First posted 2019-09-20 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2021-08

CONDITIONS: PreDiabetes
Keywords: prediabetes; TCM; body constitution; meridian energy; APP
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Routine care.
- Experimental group (Experimental): The participants accept TCM regimen-based lifestyle mobile health application intervention.
  Interventions: Other: Traditional Chinese medicine regimen-based lifestyle mobile health APP
- Sham comparator group (Sham Comparator): The participants accept mobile health application intervention.
  Interventions: Other: Lifestyle mobile health APP

INTERVENTIONS:
Other: Traditional Chinese medicine regimen-based lifestyle mobile health APP — The Experimental group receives TCM regimen-based lifestyle mobile health application intervention.
  Arms: Experimental group
Other: Lifestyle mobile health APP — Sham comparator group receives mobile health application, but there is no traditional Chinese medicine information.
  Arms: Sham comparator group

SUMMARY:
Prediabetes is a major risk factor for diabetes. The Lifestyle Modification Mobile Health Application (APP) could not only help to decrease blood sugar among individuals with prediabetes but it could also prevent a later occurrence of diabetes. While many people use traditional Chinese medicine (TCM) to improve the participants body constitution in Chinese culture, it rarely if ever obtained through a mobile device. There are very few apps that provide effective TCM regimen-based lifestyle advice for prediabetes. Therefore, the investigators want to develop and evaluate the effectiveness of receiving TCM regimen-based lifestyle advice from a mobile device designed to improve the applicant's health status.

DETAILED DESCRIPTION:
Background: People with prediabetes have an increased risk of Type 2 diabetes. Traditional Chinese medicine (TCM) lifestyle modification has been shown to be effective in achieving a balanced status and decreasing the risk of prediabetes progressing to diabetes. TCM theories note that Body constitution (BC) lays the foundation for diagnosis, treatment and disease prevention. The measurement and regulation of an individual's body constitution might prevent disease. TCM practitioners give individualized interventions according to each person's body constitution. Qi (energy) also is a core concept in TCM. Both body constitution and meridian energy (ME) can be used to determine deviated and abnormal body function. The Lifestyle Modification Mobile Health Application (APP) could help to decrease blood sugar among individuals with prediabetes, it could also prevent a later occurrence of diabetes. But, a few studies to development a TCM regimen-based lifestyle APP, and evaluate the effectiveness of receiving TCM regimen-based lifestyle APP in prediabetes. In this study, the objective was to development a TCM regimen-based lifestyle APP, and evaluate the effectiveness of receiving TCM regimen-based lifestyle APP in prediabetes.

Aims of the study: To development a TCM regimen-based lifestyle APP, and evaluate the effectiveness of receiving TCM regimen-based lifestyle APP in prediabetes.

Materials and Methods: A three-arm randomized controlled trail. The study was carried out involving 121 participants, who were recruited at a teaching hospital in northern Taiwan. The study variables include socio-demographics, disease history, and lifestyle, the blood glucose and BMI data from the blood-test will be obtained from the online medical charts. Physical activity was measured by International Physical Activity Questionnaire Self-Administered Taiwan Version. Health related quality of life was assessed by the SF-36, which yielded physical component score (PCS) and mental component scores (MCS), with higher score indicating better quality of life. The Body Constitution questionnaire (BCQ) was used to measure neutral, Yang-deficiency, Ying-deficiency, and Phlegm-stasis, with higher scores indicating larger deficiencies. Meridian energy was examined by using the Meridian energy device, which included individual meridian energy.

Possible effect: There is no TCM regimen-based lifestyle mobile health APP among people with prediabetes. Through the study, The investigators hope to develop a TCM regimen-based lifestyle mobile health APP, and evaluation it. By TCM regimen-based lifestyle using and use of APP, health management of the could be improved. The results could serve as a reference for promotion of traditional Chinese preventive medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Previously diagnosed with prediabetes with an HbA1c of 5.7% to 6.4% and an FPG level of 100 mg/dl to < 126 mg/dl (ADA, 2011, 2014).
2. Aged 20 and above.
3. Provided informed consent.

Exclusion Criteria:

1. Use of hypoglycemic agent,βblocker, thiazide diuretics, nicotinic acid or steroids within the past 3 months.
2. Self-reported catastrophic illness in the last 6 months (e.g. stroke, cardiovascular disease, renal and liver insufficiency, heart failure, chronic obstructive pulmonary disease and cancer).
3. Endocrine diseases like hyperthyroidism or autoimmune disease.
4. Psychosis or other major neurocognitive disorder; (e) pregnancy and/or lactation.

(f) Individuals with pacemakers.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Meridian energy of Meridian energy device | Change before, through intervention completion (average of 3 months)and after 1 month intervention.
  The meridian energy device captures data regarding the individual's balance of meridian energy. Balance was measured by the values of physical, metabolism, musculoskeletal and circulation, mental health, and autonomic nervous system status ratios. To achieve the appropriate balance for the energy results, a ratio of close to one was preferred.
Body constitution of body constitution questionnaire (BCQ) | Change before, through intervention completion (average of 3 months)and after 1 month intervention.
  The scale range from 44 to 220, with higher scores indicating larger deficiencies
Blood sugar control of fasting plasma glucose (FPG) | Change before, through intervention completion (average of 3 months)and after 1 month intervention.
  The normal range of FPG from 70-99mg/dL.
Blood sugar control of HbA1c | Change before, through intervention completion (average of 3 months)and after 1 month intervention.
  The normal range of HbA1c from 4-5.6%.
Health-related quality of life of short form 36 (SF-36) | Change before, through intervention completion (average of 3 months)and after 1 month intervention.
  The scale range from 0 to 100, with higher scores indicating better quality of life

SECONDARY OUTCOMES:
Physical activity of international physical activity questionnaire self-administered short version (IPAQ-SS) | Change before, through intervention completion (average of 3 months)and after 1 month intervention.
  The unit of measurement is metabolic equivalent (METs), with higher METs indicating more physical activity
Dietary behavior of the dietary behavior questionnaire | Change before, through intervention completion (average of 3 months)and after 1 month intervention.
  The scores ranged from 14 to 56, with higher scores indicating a better corresponding to the Dietary Approaches to Stop Hypertension (DASH) diet.
Body mass index (BMI) | Change before, through intervention completion (average of 3 months)and after 1 month intervention.
  The normal range of BMI from 18.5-24.9 kg/m2.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Tzu Chi Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chung HW, Tai CJ, Chang P, Su WL, Chien LY. The Effectiveness of a Traditional Chinese Medicine-Based Mobile Health App for Individuals With Prediabetes: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2023 Jun 20;11:e41099. doi: 10.2196/41099. PMID 37338977